CLINICAL TRIAL: NCT04943042
Title: An Observational, Multicenter Study to Evaluate the Use and Effectiveness of Doptelet® (Avatrombopag) in Adult Patients With Immune Thrombocytopenia (ITP)
Brief Title: An Observational, Multicenter Study to Evaluate the Use and Effectiveness of Doptelet® in Patients With ITP
Acronym: ADOPT
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Doptelet-001
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia; ITP
Keywords: TPO RA (thrombopoietin receptor agonists )
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Full-analysis set (FAS): The FAS includes all enrolled patients. The FAS will be used for all analyses.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — According to prescription
  Other Names: Doptelet®

SUMMARY:
This is a multi-center, observational, Phase 4 study in patients with Immune Thrombocytopenia (ITP) designed to describe the real-world effectiveness of Doptelet and assess the patterns of drug utilization to add to the knowledge base regarding the use of Doptelet in routine medical practice. Patients eligible for participation will, as part of their routine medical care, be receiving Doptelet for the treatment of ITP.

DETAILED DESCRIPTION:
This is a multi-center, observational, Phase 4 study in patients with ITP designed to describe the real-world effectiveness of Doptelet and assess the patterns of drug utilization to add to the knowledge base regarding the use of Doptelet in routine medical practice.

Patients eligible for participation will, as part of their routine medical care, be receiving Doptelet for the treatment of ITP.

The scope of the study is to collect both retrospective and prospective data. The main part of the study will be prospective collecting data on usage, effectiveness, safety, patient- and clinician-reported outcomes and health economic parameters whereas the retrospective part will consist of collection of information on previous treatments, reason for treatment switch, healthcare resource use and, if applicable, Doptelet treatment prior to enrollment. The retrospective data collection will be based on the information available in the patient's medical records. Data will be collected for up to 12 months prior to Doptelet treatment start.

Prospective data will be collected at routine clinical visits throughout the study. Patients will be followed for 12 (+6) months and will be enrolled until their first scheduled visit after 12 months of enrollment, or until early termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age
2. Established and well documented ITP diagnosis
3. Patient is treated with, or at enrollment prescribed, Doptelet for ITP. Decision to initiate treatment shall be made by the treating physician and independently from the decision to include the patient in the study
4. Signed and dated informed consent provided by the patient before any study-related activities are undertaken
5. Willing and able to comply with protocol requirements

Exclusion Criteria:

1. Enrollment in a concurrent clinical interventional study, or intake of an Investigational Medicinal Product (IMP), within three months prior to inclusion in this study
2. ITP secondary to Evan's syndrome, lupus and other autoimmune diseases
3. ITP secondary to other hematological disorders and hematological malignancies
4. ITP secondary to any other malignancies
5. ITP secondary to known drug toxicity
6. ITP secondary to any other disease considered relevant by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Investigators will attempt to consecutively enroll all eligible patients who present for a routine clinical visit or during a routine visit where the patient is started on Doptelet treatment (new users of Doptelet).
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Cumulative number of weeks with a platelet count ≥30×109/L during Doptelet treatment. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Laboratory measures of platelet count will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts will be based on local laboratory results. Platelet count is an accepted surrogate marker for bleeding risk. Platelet count is a standard measurement commonly used both in clinical practice and in studies in patients with ITP.
  Platelet counts during rescue medication use and within 4 weeks after stopping a rescue medication or following splenectomy will not be counted in the cumulative number of weeks.

SECONDARY OUTCOMES:
Cumulative number of weeks with a platelet count ≥50×109/L during Doptelet treatment. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Laboratory measures of platelet count will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts will be based on local laboratory results. Platelet count is an accepted surrogate marker for bleeding risk. Platelet count is a standard measurement commonly used both in clinical practice and in studies in patients with ITP.
  Platelet counts during rescue medication use and within 4 weeks after stopping a rescue medication or following splenectomy will not be counted in the cumulative number of weeks.
Number and proportion of patients with a platelet count ≥30×109/L, for at least 8 consecutive weeks. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Laboratory measures of platelet count will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts will be based on local laboratory results.Platelet count is an accepted surrogate marker for bleeding risk. Platelet count is a standard measurement commonly used both in clinical practice and in studies in patients with ITP.
Number and proportion of patients with a platelet count ≥50×109/L for at least 8 consecutive weeks. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Laboratory measures of platelet count will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts will be based on local laboratory results.Platelet count is an accepted surrogate marker for bleeding risk. Platelet count is a standard measurement commonly used both in clinical practice and in studies in patients with ITP.
Number and proportion of patients experiencing WHO bleeding grade ≥ 2. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  All bleeding events will be assessed by the Investigator according to the WHO bleeding scale where the severity of the bleeding is graded from 0 to 4 (0=no bleeding; 1=petechial bleeding; 2=mild blood loss (clinically significant); 3=gross blood loss; requires transfusion (severe); 4=debilitating blood loss, retinal or cerebral associated with fatality).
Number and proportion of patients requiring rescue medication. | Data will be collected retrospectively via the medical records for a time period of 12 months prior to Doptelet start as well as prospectively for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via the patient's medical records.
Time from Doptelet treatment start to platelet count ≥30×109/L. | Data will be collected retrospectively via the medical records for a time period of 12 months prior to Doptelet start as well as prospectively for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Laboratory measures of platelet count will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts will be based on local laboratory results.Platelet count is an accepted surrogate marker for bleeding risk. Platelet count is a standard measurement commonly used both in clinical practice and in studies in patients with ITP.
Time from Doptelet treatment start to platelet count ≥50×109/L. | Data will be collected retrospectively via the medical records for a time period of 12 months prior to Doptelet start as well as prospectively for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Laboratory measures of platelet count will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts will be based on local laboratory results.Platelet count is an accepted surrogate marker for bleeding risk. Platelet count is a standard measurement commonly used both in clinical practice and in studies in patients with ITP.
Doptelet dose and dosing frequency per patient (assessed by prescription). | Data will be collected retrospectively via the medical records for a time period of 12 months prior to Doptelet start as well as prospectively for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via the patient's medical records.
Adherence to Doptelet treatment assessed via the 8-item Morisky Medication Adherence Scale (MMAS-8). | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  MMAS-8 is an 8-item structured, self-reported medication adherence measure. The self-reported measure of medication taking was developed from a previously validated 4-item scale and supplemented with additional items addressing the circumstances surrounding adherence behavior. Each item measures a specific medication-taking behavior and not a determinant of adherence behavior. Response categories are yes/no for each item with a dichotomous response and a 5-point Likert response for the last item. Adherent patients are identified with the score of 8 on the scale, medium adherers with a score of 6 to <8, and low adherers with a score of <6.
  The MMAS-8 Scale, content, name, and trademarks are protected by US copyright and trademark laws. Permission for use of the scale and its coding is required. A license agreement is available from Donald E. Morisky, ScD, ScM, MSPH; donald.morisky@moriskyscale.com.
Reason for ITP treatment discontinuation or change from one ITP treatment to another, prior to as well as during the study. | Data will be collected retrospectively via the medical records for a time period of 12 months prior to Doptelet start as well as prospectively for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via the patient's medical records.
Patient satisfaction with outcome of Doptelet treatment using the Treatment Satisfaction Questionnaire for Medication (TSQM-9). | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  TSQM-9 is a self-administered generic measure to assess patients' satisfaction with their medication. It consists of nine items distributed across three dimensions: Effectiveness (3 items), Convenience (3 items) and Global satisfaction scale (3 items). Each domain score ranges from 0 to 100, higher score indicating greater satisfaction.
Physician satisfaction with outcome of Doptelet treatment using a 5 point scale. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  The treating physician will evaluate satisfaction with the Doptelet treatment by answering the question: "On a scale of 1-5 with 5 being highly satisfied and 1 being highly dissatisfied, how would you rate your satisfaction with the desired treatment outcome of the Doptelet treatment?"
Physician assessment of clinical change of Doptelet treatment using the Clinical Global Impression of Change (CGIC) scale. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  The treating physician will evaluate the clinical change of Doptelet treatment by grading the change on a 7-point scale; very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Change from enrollment in the European Quality of Life - 5 Dimensions (EQ-5D-5L) scale. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  The EQ-5D is a standardized generic instrument for use as a measure of health outcome. The EQ-5D consists of 2 parts - the EQ-5D descriptive profile which is mapped into a single index value for health status (utility value) and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Change from enrollment in the Immune Thrombocytopenic Purpura Patient Assessment Questionnaire (ITP-PAQ). | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  ITP-PAQ is a disease-specific self-administered tool which was developed and validated to assess health related quality of life (HRQoL) in adult patients with ITP using a 4-week recall period. It consists in 44 items distributed across 10 dimensions: Symptoms (6 items), Bother-Physical Health (3 items), Fatigue/Sleep (4 items), Activity (2 items), Fear (5 items), Psychological Health (5 items), Work (4 items), Social Activity (4 items), Women's Reproductive Health (6 items) and Overall QoL (5 items). Each scale is scored from 0 to 100, with higher scores representing better HRQoL.
Change from enrollment in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) questionnaire. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  FACIT-Fatigue is a 13-item scale developed to assess specifically quality of life concerns related to fatigue in patients with chronic diseases. The scale was initially developed to assess cancer-related fatigue, however it has been since then used and psychometrically validated in other chronic diseases, including ITP. The instrument includes items such as tiredness, weakness, listlessness, lack of energy, and the impact of these feelings on daily functioning over the past seven days. Each item is scored on a 5-point Likert Scale ranging from "0-Not at all" to "4-Very much".
Change from enrollment in Patient Global Impression of Change (PGIC) scale. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  PGIC will be used to evaluate patients' perception of changes in the severity of their ITP symptoms on the scale: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Change from enrollment in Work Productivity and Activity Impairment (WPAI) questionnaire. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  WPAI for specific health problem, WPAI:SHP v2.0 questionnaire is a generic and standard instrument developed to measure the effect of specific health problems and symptom severity on work productivity and regular activities during the past seven days. It contains six items which ascertain employment status and quantify absenteeism due to health problems, presenteeism and overall health-related impairment in both paid work and regular activities over the previous 7 days. The WPAI provides quantitative data at the item level compatible with economic modelling.
Healthcare resource use including; Inpatient and /or outpatient visits since last routine visit. | Data will be collected retrospectively via the medical records for a time period of 12 months prior to Doptelet start as well as prospectively for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  The following data related to in-patient and/or out-patient visits since last routine visit will be collected:
  * Length of hospitalization
  * Reason for visit
  * Surgical procedures
  * ICU stay, CT scans
  * Regular blood tests and haemato-chemistry blood tests
  * Platelet transfusions
  * Other.
Use of concomitant ITP medications throughout the study. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via the patient's medical records.
Serious adverse events (SAEs) | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via reports from the Investigators based on the patient's medical records.
Adverse events of special interest (AESIs) (e.g., thromboembolic events, significant bleeding (WHO bleeding scale grade ≥ 3)). | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via reports from the Investigators based on the patient's medical records.
AEs leading to Doptelet discontinuation. | Data will be collected for all routine visits completed during the study period which is at least 12 but not more than 18 months.
  Information will be collected via reports from the Investigators based on the patient's medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Skuban, MD, Study Director — Swedish Orphan Biovitrum AB; Vickie McDonald, MD, Study Director — Royal London Hospital, London, UK
Locations (55):
- Swedish Orphan Biovitrum Research Site 131, Zagreb, Croatia
- Czechia (5):
  - Swedish Orphan Biovitrum Research Site 122, Brno
  - Swedish Orphan Biovitrum Research Site 123, Ostrava
  - Swedish Orphan Biovitrum Research Site 121, Prague
  - Swedish Orphan Biovitrum Research Site 124, Prague
  - Swedish Orphan Biovitrum Research Site 125, Prague
- Germany (14):
  - Swedish Orphan Biovitrum Research Site 108, Aschaffenburg
  - Swedish Orphan Biovitrum Research Site 114, Augsburg
  - Swedish Orphan Biovitrum Research Site 116, Augsburg
  - Swedish Orphan Biovitrum Research Site 103, Bad Homburg
  - Swedish Orphan Biovitrum Research Site 106, Berlin
  - Swedish Orphan Biovitrum Research Site 113, Dresden
  - Swedish Orphan Biovitrum Research Site 102, Frankfurt
  - Swedish Orphan Biovitrum Research Site 105, Frankfurt
  - Swedish Orphan Biovitrum Research Site 104, Hanover
  - Swedish Orphan Biovitrum Research Site 112, Kaiserslautern
  - Swedish Orphan Biovitrum Research Site 101, Kassel
  - Swedish Orphan Biovitrum Research Site 115, Leipzig
  - Swedish Orphan Biovitrum Research Site 109, Schorndorf
  - Swedish Orphan Biovitrum Research Site 111, Stolberg
- Italy (8):
  - Swedish Orphan Biovitrum Research Site 509, Bologna
  - Swedish Orphan Biovitrum Research Site 504, Catania
  - Swedish Orphan Biovitrum Research Site 502, Florence
  - Swedish Orphan Biovitrum Research Site 506, Meldola
  - Swedish Orphan Biovitrum Research Site 511, Milan
  - Swedish Orphan Biovitrum Research Site 510, Milan
  - Swedish Orphan Biovitrum Research Site 503, Roma
  - Swedish Orphan Biovitrum Research Site 505, Rome
- Netherlands (3):
  - Swedish Orphan Biovitrum Research Site 202, Apeldoorn
  - Swedish Orphan Biovitrum Research Site 204, Arnhem
  - Swedish Orphan Biovitrum Research Site 203, The Hague
- Norway (2):
  - Swedish Orphan Biovitrum Research Site 302, Bergen
  - Swedish Orphan Biovitrum Research Site 301, Oslo
- Spain (11):
  - Swedish Orphan Biovitrum Research Site 611, Barcelona
  - Swedish Orphan Biovitrum Research Site 609, Burgos
  - Swedish Orphan Biovitrum Research Site 610, Granada
  - Swedish Orphan Biovitrum Research Site 601, Madrid
  - Swedish Orphan Biovitrum Research Site 605, Madrid
  - Swedish Orphan Biovitrum Research Site 607, Murcia
  - Swedish Orphan Biovitrum Research Site 606, Oviedo
  - Swedish Orphan Biovitrum Research Site 608, Palma de Mallorca
  - Swedish Orphan Biovitrum Research Site 602, Salamanca
  - Swedish Orphan Biovitrum Research Site 604, Seville
  - Swedish Orphan Biovitrum Research Site 603, Vigo
- Switzerland (2):
  - Swedish Orphan Biovitrum Research Site 802, Basel
  - Swedish Orphan Biovitrum Research Site 801, Lausanne
- United Kingdom (9):
  - Swedish Orphan Biovitrum Research Site 709, Edinburgh, Scotland
  - Swedish Orphan Biovitrum Research Site 708, Glasgow, Scotland
  - Swedish Orphan Biovitrum Research Site 701, Bristol
  - Swedish Orphan Biovitrum Research Site 704, Leicester
  - Swedish Orphan Biovitrum Research Site 707, London
  - Swedish Orphan Biovitrum Research Site 710, London
  - Swedish Orphan Biovitrum Research Site 705, Newcastle
  - Swedish Orphan Biovitrum Research Site 702, Nottingham
  - Swedish Orphan Biovitrum Research Site 703, Oxford

IPD SHARING:
Plan to Share IPD: Yes
According to Sobi's data sharing policy Sobi may share anonymized clinical study data with qualified researchers. Sobi commits to sharing clinical study data on participant level and summary data for medicines and indications approved by the European Medicines Agency (EMA) and/or the Food and Drug Administration (FDA). Data access will be granted in response to qualified research requests. All requests are evaluated by a cross functional panel of experts within Sobi.
Time Frame: Evaluated on a case by case basis
Access Criteria: A decision on data sharing will be based on the following:
  * The scientific merit of the proposal - i.e. the proposal should be scientifically sound, ethical, and have the potential to contribute to the advancement of public health.
  * The feasibility of the research proposal - i.e. the requesting research team must be scientifically qualified and have the resources to conduct the proposed project.
  * Maintenance of personal integrity - i.e. Sobi will not consider sharing individual data if there is a risk of re-identification of individuals despite a proper anonymisation. Moreover, the patients' informed consent will always be respected. Sobi reserves the right to reject the proposal if the anonymisation process will render unusable data.
  * Publication of results - the applicants should commit to submit their findings to a peer-reviewed scientific journal, alternatively to present the results at a congress (poster or similar), regardless of the research outcome.
URL: https://www.sobi.com/en/policies